CLINICAL TRIAL: NCT06809790
Title: The Effect of Dry Needling of the Upper Trapezius Muscle Added to Therapeutic Exercise Therapy on the Thickness of the Cervical Muscles in Myofascial Pain Syndrome
Brief Title: Dry Needling Combined With a Therapeutic Exercise Program in Myofascial Pain Syndrome: Sonographic Evaluation of Cervical Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammed Oğuz, Medical Doctor, Istanbul Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18/09/2024;2024-KAEK-30;114
Record Dates: First submitted 2025-01-26; First posted 2025-02-05 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Myofascial Pain Syndrome - Neck; Myofascial Pain of Upper Trapezius Muscle
Keywords: myofascial pain syndrome; trigger point; dry needling; upper trapezius muscle; Therapeutic Exercise
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into two groups; the first group will receive only exercise therapy, and the second group will receive exercise therapy as well as dry needling treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Therapeutic Exercise (Active Comparator)
  Interventions: Behavioral: Therapeutic Exercise Program
- Group 2: Therapeutic Exercise and Dry Needling (Active Comparator)
  Interventions: Behavioral: Therapeutic Exercise Program; Procedure: Dry Needling

INTERVENTIONS:
Behavioral: Therapeutic Exercise Program — Participants in this group will receive a therapeutic exercise program (including cervical range of motion and trapezius stretching) during the study period.
Procedure: Dry Needling — Participants in this group will receive dry needling treatment for active trigger points in addition to the therapeutic exercise program. Dry needling treatment will be applied in a total of 3 sessions at 0, 1, and 2. weeks, one week apart.
  Arms: Group 2: Therapeutic Exercise and Dry Needling

SUMMARY:
Patients between the ages of 20-65 years who present to the Physical Medicine and Rehabilitation outpatient clinics of our hospital with complaints of back and neck pain and are diagnosed with myofascial pain syndrome will be referred to the physicians responsible for the study to be included in the study. Exclusion criteria will be reviewed, and patients with chronic pain for more than 3 months and an active trigger point in the unilateral upper trapezius muscle will be included in the study. Patients will be randomly divided into two groups; the first group will receive only exercise therapy (including cervical range of motion and trapezius stretching), and the second group will receive exercise and dry needling therapy (1 time per week, 3 sessions in total). Demographic data (age, gender, body mass index, occupation) of all patients included in the study will be recorded. The relationship between pain and loss of function according to the Visual Analog Scale (VAS), Short Form 36 (SF-36), and Neck Disability Index (NDI) scales will be recorded. Bilateral upper trapezius, sternocleidomastoideus, and total cervical extensor muscle thickness (upper trapezius, splenius capitis, semispinalis capitis, semispinalis cervicis, and multifidus) and longus colli muscle thickness measurements will be made with the ultrasonography device in our clinic. The first group will receive only exercise therapy after the measurements. Patients in the second group will receive a total of 3 sessions of dry needling treatment to the trapezius muscle for active trigger points at 0, 1, and 2 weeks in addition to exercise therapy. After the initial examination, control VAS, SF-36, NDI, and control ultrasonographic measurements will be performed in all patients at the 3rd week and 6th week. Using data analysis methods, the effect of dry needling treatment for active trigger points in the trapezius muscle on pain and functionality as well as the thickness of the cervical muscles will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-65 years with neck pain for more than 12 weeks
* Active trigger point in the unilateral upper trapezius muscle on physical examination
* Who agreed not to receive anti-inflammatory and myorelaxant treatment during the study period

Exclusion Criteria:

* Patients diagnosed with rheumatologic diseases
* Patients with radiculopathy
* Patients with a history of previous surgery in the shoulder, back, and neck region
* Patients with polyneuropathy
* Patients with severe cervical spondylosis
* Patients with cerebrovascular events
* Patients with malignancies
* Those with cognitive impairment
* Those with bleeding disorders
* Patients diagnosed with fibromyalgia
* Patients with thyroidectomy
* Anti-inflammatory-analgesic or myorelaxant treatment within the last 1 month
* Patients with a history of injection into the upper trapezius muscle or cervical region within the last 3 months

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2025-02-09 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic evaluation for muscle thickness assessment | It will be evaluated in the baseline, third, and sixth weeks.
  Bilateral upper trapezius, sternocleidomastoid, total cervical extensor muscle thickness (upper trapezius, splenius capitis, semispinalis capitis, semispinalis cervicis, and multifidus), and longus colli muscle thickness measurements will be made with the ultrasonography device.

SECONDARY OUTCOMES:
Pain will be assessed with Visual Analog Scale. | It will be evaluated in the baseline, third, and sixth weeks.
  Visual Analog Scale (VAS) score ranges from 0 to 10. High scores describe more pain, and low scores describe less pain.
Functional status will be assessed with the Neck Disability Index. | It will be evaluated in the baseline, third, and sixth weeks.
  Neck Disability Index (NDI) consists of 10 questions in total. Each question receives a score ranging from 0 to 5. Totals can have a minimum score of 0 and a maximum score of 50. Higher scores indicate more severe disability.
General health status will be assessed with Short Form 36. | It will be evaluated in the baseline, third, and sixth weeks.
  Short Form 36 (SF-36) is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Oğuz, Principal Investigator — Istanbul Training and Research Hospital
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Fatih, Turkey (Türkiye)